CLINICAL TRIAL: NCT04219241
Title: Clinical Extension Study for Assessing the Safety and Efficacy of the Intravenous Administration of Cellavita-HD in Huntington's Disease Patients Who Participated in the ADORE-DH Study.
Brief Title: Clinical Extension Study for Safety and Efficacy Evaluation of Cellavita-HD Administration in Huntington's Patients.
Acronym: ADORE-EXT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azidus Brasil (Industry)
Collaborators: Cellavita Pesquisa Científica Ltda (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADORE-EXT; 23917319.0.0000.5412 (Registry Identifier: CAAE)
Record Dates: First submitted 2019-12-11; First posted 2020-01-07 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Huntington Disease
Keywords: Huntington Disease; Stem cell therapy; Dental Pulp Stem Cell
MeSH Terms: conditions — Huntington Disease | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cellavita-HD (Experimental): The participants will receive a total of 12 intravenous administrations of 2x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 180 days (total of 4 cycles).
  Interventions: Biological: Cellavita-HD

INTERVENTIONS:
Biological: Cellavita-HD — The participants will receive a total of 12 intravenous administrations of 2x10^6 cells/weight range divided into three administrations per cycle. Each administration will occur every 30 days and cycles every 180 days (total of 4 cycles).
  Other Names: cellular therapy, mesenchymal stem cells

SUMMARY:
Cellavita-HD is a stem-cell therapy for Huntington's Disease. Open label, single treatment, extension study for long-term safety and efficacy evaluation of Cellavita-HD intravenous administration in Huntington's disease patients who participated of ADORE-DH trial.

DETAILED DESCRIPTION:
This extension study will include the subjects who participated the study phase II for dose-response evaluation of Cellavita-HD intravenous administration in Huntington's disease patients (maximum 35 subjects). Because it is a extension study, with an open scenario, the subjects will receive the maximum dose tested in the last clinical trial (ADORE-DH), corresponding to 6 x 10^6 cells/weight range for each treatment cycle planned. Throughout of 24 months, the subjects will receive total dose planned divided into three administrations per cycle (2 x 10^6 cells/weight range), that each will occur every 30 days. The maintaining the effectiveness of intravenous administration of Cellavita-HD product over time on clinical progression Huntington's disease will be verified by comparing the UHDRS total score at the end of the 24th study month against baseline score. Secondary evidences of efficacy will be evaluated by through the data of functional state, total functional capacity, functional independence, psychiatric symptoms and cognition from UHDRS scale. Additionally, related data to clinical worsening, change of Body Mass Index (BMI), risk of suicide attempt and neurological image improvement will be evaluated. Safety evaluation will included the incidence and classification of the adverse events experienced by the subjects during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Phase II study participants (ADORE-DH) who express interest in participating in the extension period and who may have significant clinical benefits (motor, cognitive, behavioral and functional capacity) at the Investigator's judged after intravenous application of the Cellavita-HD product;
2. Provide consent by signing in two copies of the Informed Consent Form;
3. Participant using an acceptable contraceptive method.

Exclusion Criteria:

1. History of malignant neoplasia;
2. Present any clinical and laboratory condition or comorbidity that, at the physician's judged, may endanger the health of the research participant and prevent him / her from being part of the extension study;
3. known hypersensitivity to the investigational product and / or products of bovine origin;
4. Research participant who has participated in clinical trial protocols in the last twelve (12) months, unless the Investigator believes that there may be direct benefit to it (Resolution CNS 251 of August 7, 1997, item III, sub-item J);
5. Pregnant or lactating participant;
6. In use or anticipated use of immunosuppressive drugs as well as any other drug in which the use is restricted to this research protocol.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-02-10 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Maintenance of effectiveness on clinical progression of the disease | Two years (every study visit)
  The maintenance of treatment effectiveness will be verified by comparing the total UHDRS (Unified Huntington's Disease Rating Scale) score registered at the end of the 24th month of study in relation to the baseline score.

SECONDARY OUTCOMES:
Clinical neurological worsening over the treatment by UHDRS | Two years
  The clinical neurological worsening over the treatment will be evaluated by specific Unified Huntington's Disease Rating Scale - UHDRS subscales (motor, behavior, functional capacity and cognitive domain). Each specific domain have 4 categories (from 0 to 4). For motor subscale, the score ranged from 0 to 124; Therefore,highest scores indicate more severe motor impairment. Cognitive operations are assessed by aplication of three tests: verbal fluency test, Symbol Digit modalities test and the Stroop Color Word test. For all cognitive tests, highest scores translate to better cognitive ability. Behavior assessment score is obtained by summing different items related to the severity of psychiatric symptoms. Highest scores indicate greater behavioral impairment. Functional assessment includes three scales: a functional checklist, an independence scale, and a total functional capacity assessment. The maximum score of 25 points represents greater functional capacity.
BMI assessment | Two years
  The BMI (Body Mass Index) will be evaluated through the BMI profiles obtained during the treatment to evaluate the nutritional status.
Risk of suicidal ideation and/or behavior by C-SSRS | Two years
  Will be evaluated by Columbia Suicide Severity Rating Scale (C-SSRS) registered throughout the study in relation to the baseline score. The total score ranges from 2 to 25, with a higher number indicating more intense ideation and greater risk. Greater lethality or potential lethality of the behavior (endorsed on the Behavior subscale) indicates increased risk.
Risk of suicidal ideation and/or behavior by HDS | Two years
  Will be evaluated through Suicidal Domain from HDS (Hamilton Depression Scale) registered throughout the study in relation to the baseline score. Scores above 25 points characterize severely ill patients depressed; scores between 18 and 24 points, moderately depressed patients; and scores between 7 and 17 points, patients with mild depression.
CNS assessment by MRI (Magnetic Ressonance Imaging) | One year
  Huntington's patients normally present MRI structural abnormalities, including cortical atrophy and structural white matter changes. Alterations after product administration will be evaluated througout statistical comparison of the CNS assessment through magnetic resonance imaging at cortical thickness measurements, volumes of different brain structures, especially the basal ganglia, with special attention to caudate and metabolic changes identified in proton spectroscopy.

OTHER OUTCOMES:
Safety of Cellavita-HD administration | Two years
  Will be evaluated from the periodical assessments including clinical and imaging exams. Any clinical relevant change will be properly recorded and judged by Investigator according to expectation, causality, intesity and severity, as well as the continued treatment administration.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Macedo, MD, Principal Investigator — Azidus Brasil Scientific Research and Development Ltda
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
It is believed that after the data analysis and presentation to the National Commission on Research Ethics, all data will become public.

REFERENCES:
- [Background] Adachi N, Numakawa T, Richards M, Nakajima S, Kunugi H. New insight in expression, transport, and secretion of brain-derived neurotrophic factor: Implications in brain-related diseases. World J Biol Chem. 2014 Nov 26;5(4):409-28. doi: 10.4331/wjbc.v5.i4.409. PMID 25426265
- [Background] Aleynik A, Gernavage KM, Mourad YSh, Sherman LS, Liu K, Gubenko YA, Rameshwar P. Stem cell delivery of therapies for brain disorders. Clin Transl Med. 2014 Jul 19;3:24. doi: 10.1186/2001-1326-3-24. eCollection 2014. PMID 25097727
- [Background] Bachoud-Levi AC, Gaura V, Brugieres P, Lefaucheur JP, Boisse MF, Maison P, Baudic S, Ribeiro MJ, Bourdet C, Remy P, Cesaro P, Hantraye P, Peschanski M. Effect of fetal neural transplants in patients with Huntington's disease 6 years after surgery: a long-term follow-up study. Lancet Neurol. 2006 Apr;5(4):303-9. doi: 10.1016/S1474-4422(06)70381-7. PMID 16545746
- [Background] Barker RA, Mason SL, Harrower TP, Swain RA, Ho AK, Sahakian BJ, Mathur R, Elneil S, Thornton S, Hurrelbrink C, Armstrong RJ, Tyers P, Smith E, Carpenter A, Piccini P, Tai YF, Brooks DJ, Pavese N, Watts C, Pickard JD, Rosser AE, Dunnett SB; NEST-UK collaboration. The long-term safety and efficacy of bilateral transplantation of human fetal striatal tissue in patients with mild to moderate Huntington's disease. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):657-65. doi: 10.1136/jnnp-2012-302441. Epub 2013 Jan 23. PMID 23345280
- [Background] Goldberg YP, Kremer B, Andrew SE, Theilmann J, Graham RK, Squitieri F, Telenius H, Adam S, Sajoo A, Starr E, et al. Molecular analysis of new mutations for Huntington's disease: intermediate alleles and sex of origin effects. Nat Genet. 1993 Oct;5(2):174-9. doi: 10.1038/ng1093-174. PMID 8252043
- [Background] Unified Huntington's Disease Rating Scale: reliability and consistency. Huntington Study Group. Mov Disord. 1996 Mar;11(2):136-42. doi: 10.1002/mds.870110204. PMID 8684382
- [Background] Jia JM, Chen Q, Zhou Y, Miao S, Zheng J, Zhang C, Xiong ZQ. Brain-derived neurotrophic factor-tropomyosin-related kinase B signaling contributes to activity-dependent changes in synaptic proteins. J Biol Chem. 2008 Jul 25;283(30):21242-50. doi: 10.1074/jbc.M800282200. Epub 2008 May 12. PMID 18474605
- [Background] Kerkis I, Haddad MS, Valverde CW, Glosman S. Neural and mesenchymal stem cells in animal models of Huntington's disease: past experiences and future challenges. Stem Cell Res Ther. 2015 Dec 14;6:232. doi: 10.1186/s13287-015-0248-1. PMID 26667114
- [Background] Marder K, Zhao H, Myers RH, Cudkowicz M, Kayson E, Kieburtz K, Orme C, Paulsen J, Penney JB Jr, Siemers E, Shoulson I. Rate of functional decline in Huntington's disease. Huntington Study Group. Neurology. 2000 Jan 25;54(2):452-8. doi: 10.1212/wnl.54.2.452. PMID 10668713